CLINICAL TRIAL: NCT07269821
Title: Evaluation of a Nutritional Intervention With Dietary Supplements in People Who Have Recently Lost Weight: Effects on Body Composition, Emotional Health, and Gut Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alicante (Other)
Responsible Party: Principal Investigator, Prof. Dr. Alejandro Martínez-Rodríguez, Catedrático Ciencias de la Salud, University of Alicante
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UA-2025-05-22_2
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: GLP-1; Weight Loss Trajectory; Emotional Disorder; Microbiota Balance
Keywords: weight loss maintenance; GLP-1 receptor agonists; body composition; fat-free mass; nutritional supplementation; polyphenols; prebiotics; gut microbiota; emotional well-being; metabolic recovery; post-weight-loss intervention; nutraceuticals
MeSH Terms: conditions — Body-Weight Trajectory

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Experimental - Dietary supplement (Experimental): Participants will receive a daily dose of a nutraceutical formulation designed to support weight maintenance and metabolic recovery after weight loss.
  The supplement contains Metabolaid® (a standardized extract of Hibiscus sabdariffa and Lippia citriodora) aimed at improving gut microbiota composition, emotional well-being, and preserving fat-free mass.
  The intervention lasts 12 weeks, with two capsules per day, taken with meals.
  Interventions: Dietary Supplement: Metabolaid®-based nutraceutical formulation
- Arm 2: Placebo - Control (Placebo Comparator): Participants will receive a placebo identical in appearance, taste, and packaging to the active supplement.
  The placebo capsules contain inert excipients without active ingredients.
  Interventions: Dietary Supplement: Placebo capsules

INTERVENTIONS:
Dietary Supplement: Metabolaid®-based nutraceutical formulation — A 12-week supplementation with Metabolaid® to assess changes in body composition, emotional health, and gut microbiota after weight loss.
  Arms: Arm 1: Experimental - Dietary supplement
Dietary Supplement: Placebo capsules — A 12-week placebo supplementation with capsules identical in appearance to the experimental product, to evaluate differences in body composition, gut microbiota, and emotional parameters.
  Arms: Arm 2: Placebo - Control

SUMMARY:
This study aims to evaluate the effects of a 12-week nutritional intervention with dietary supplements on individuals who have experienced significant weight loss following the use of GLP-1 receptor agonists or similar weight-loss treatments. The study will investigate whether the combined supplementation protocol can improve body composition, emotional well-being, and gut microbiota diversity after discontinuation of pharmacological treatment.

Participants will be randomly assigned to one of two groups: an intervention group receiving a daily combination of food supplements containing bioactive compounds (including polyphenols, prebiotics, and antioxidants) and a placebo group. Both groups will maintain their habitual diet and lifestyle throughout the study.

Primary outcomes include changes in fat-free mass, emotional state, and gut microbiota composition. Secondary outcomes include metabolic markers, appetite regulation, and quality of life indicators.

This project seeks to provide evidence-based strategies for maintaining health and preventing metabolic rebound following rapid weight loss or pharmacologically induced appetite suppression.

DETAILED DESCRIPTION:
The increasing use of GLP-1 receptor agonists and similar drugs has led to significant weight loss in many individuals; however, this is often followed by loss of lean mass, mood alterations, and gut microbiota imbalance. This study explores a nutritional supplementation strategy designed to support metabolic recovery and preserve physiological homeostasis in this population.

This 12-week randomized, double-blind, placebo-controlled clinical trial will include adults aged 25-60 years who have recently lost ≥5% of body weight due to pharmacological treatment or restrictive dietary patterns. Participants will be randomly assigned to one of two groups:

1. Experimental Group: Daily intake of a multi-component dietary supplement containing polyphenols, prebiotic fibers, and natural extracts with antioxidant and anti-inflammatory properties.
2. Placebo Group: Daily intake of an inert product with identical appearance, taste, and packaging.

All participants will continue their usual dietary and lifestyle habits. Compliance will be monitored through periodic visits and digital tracking.

Measurements will be taken at baseline and after 12 weeks, including:

* Body composition: fat mass, fat-free mass, and phase angle.
* Blood biomarkers: glucose, lipids, liver enzymes, and inflammatory markers.
* Psychological parameters: mood, anxiety, and quality of life scales.
* Gut microbiota: analysis of microbial diversity and composition from stool samples.

The expected outcome is that the supplement will mitigate lean mass loss, improve emotional balance, and restore microbiota diversity after significant weight reduction. Results from this study may contribute to developing safe and effective strategies for post-weight-loss management and metabolic health maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 25 to 60 years.
* Documented unintentional or pharmacologically induced weight loss of ≥5% during the previous 3 months.
* Stable body weight (±2 kg variation) during the 2 weeks prior to enrollment.
* Completion or discontinuation of GLP-1 receptor agonist or other pharmacological weight-loss therapy within the last 3 months.
* Willingness to maintain habitual dietary and physical activity habits throughout the study.
* Ability to provide written informed consent and comply with all study procedures.

Exclusion Criteria:

* Current or recent use (within 3 months) of antibiotics, probiotics, or prebiotic supplements.
* Active gastrointestinal disorders (e.g., inflammatory bowel disease, celiac disease, chronic diarrhea, or severe constipation).
* Diagnosis of diabetes mellitus, cardiovascular disease, cancer, liver, or kidney dysfunction.
* Pregnancy, breastfeeding, or intention to become pregnant during the study period.
* Psychiatric disorders or use of medications affecting mood or appetite.
* Participation in another clinical trial during the previous 3 months.
* Any condition that, in the investigator's opinion, could interfere with study participation or interpretation of results.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Fat Mass (%) | Baseline and Week 12
  To evaluate changes in total fat mass percentage after the 12-week intervention, assessed by bioimpedance analysis (BIODY XPERT ZM).

SECONDARY OUTCOMES:
Change in Lean Mass (%) | Baseline and Week 12
  To evaluate changes in total lean body mass percentage after the 12-week intervention, measured by bioimpedance analysis.
Change in Visceral Fat Level | Baseline and Week 12
  To assess differences in visceral adiposity index obtained from bioimpedance measurements before and after supplementation.
Change in Body Weight (kg) | Baseline and Week 12
  To evaluate changes in body weight following the 12-week supplementation period.
Change in BMI (kg/m²) | Baseline and Week 12
  To assess changes in body mass index calculated as weight (kg) divided by height squared (m²).
Change in Waist Circumference (cm) | Baseline and Week 12
  To measure changes in abdominal circumference as an indicator of central adiposity.
Change in Hip Circumference (cm) | Baseline and Week 12
  To record changes in hip circumference to calculate waist-to-hip ratio.
Change in Gut Microbiota Diversity | Baseline and Week 12
  To evaluate changes in microbial alpha and beta diversity using 16S rRNA sequencing of stool samples.
Change in Abundance of Key Gut Microbial Taxa | Baseline and Week 12
  To analyze specific bacterial taxa abundance associated with metabolic health before and after the intervention.
Change in Appetite Score (VAS) | Baseline and Week 12
  Description: Appetite perception will be evaluated using a Visual Analogue Scale (VAS) consisting of a 100-mm horizontal line, where 0 represents "no appetite at all" and 100 represents "extremely high appetite." Participants will mark their perceived level of appetite on the line, and the score will be measured in millimeters from the left end. Range: 0-100 mm. Interpretation: Higher scores indicate greater appetite perception.
Change in Satiety Score (VAS) | Baseline and Week 12
  Description: Perceived fullness or satiety will be evaluated using a Visual Analogue Scale (VAS) consisting of a 100-mm horizontal line, where 0 represents "not at all full" and 100 represents "extremely full." Participants will indicate their perceived level of satiety on the line, and the score will be measured in millimeters from the left end. Range: 0-100 mm. Interpretation: Higher scores indicate greater perceived satiety.
Change in Physical Activity Level (IPAQ Total Score) | Baseline and Week 12
  Description: Physical activity levels will be assessed using the International Physical Activity Questionnaire - Short Form (IPAQ-SF), which records activity performed over the previous 7 days. The questionnaire includes 7 items covering walking, moderate, and vigorous activities. The total score is expressed in MET-minutes per week and categorized into low, moderate, or high activity levels. Range: 0 to unlimited MET-min/week. Interpretation: Higher scores indicate greater physical activity levels.
Change in Total Energy Intake (kcal/day) | Baseline and Week 12
  To quantify changes in daily energy consumption from dietary recalls.
Change in Macronutrient Distribution (%) | Baseline and Week 12
  To evaluate changes in carbohydrate, protein, and fat intake percentages.
Change in Fasting Glucose (mg/dL) | Baseline and Week 12
  To assess changes in fasting blood glucose levels as a metabolic indicator.
Change in Fasting Insulin (µU/mL) | Baseline and Week 12
  To measure insulin levels to assess metabolic response to supplementation.
Change in Total Cholesterol (mg/dL) | Baseline and Week 12
  To measure total cholesterol concentration in fasting blood samples.
Change in HDL Cholesterol (mg/dL) | Baseline and Week 12
  To assess HDL cholesterol changes after supplementation.
Change in LDL Cholesterol (mg/dL) | Baseline and Week 12
  To evaluate low-density lipoprotein cholesterol levels before and after intervention.
Change in Triglycerides (mg/dL) | Baseline and Week 12
  To determine the impact of supplementation on triglyceride concentrations.
Change in C-Reactive Protein (mg/L) | Baseline and Week 12
  To assess systemic inflammation through C-reactive protein levels.
Change in Interleukin-6 (pg/mL) | Baseline and Week 12
  To evaluate inflammatory status through IL-6 concentrations
Change in TNF-alpha (pg/mL) | Baseline and Week 12
  To measure tumor necrosis factor-alpha as an additional inflammatory marker

CONTACTS AND LOCATIONS:
Locations (1):
- European Institute Of Exercise and Health, Elche, Alicante, Spain